CLINICAL TRIAL: NCT02728674
Title: Management of Patients With Respiratory Symptoms in Sweden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Ekström, MD, PhD, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CASE2016
Record Dates: First submitted 2016-03-24; First posted 2016-04-05 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Breathlessness; Symptom; Opioids; Gender bias
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Sexism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Man+Breathlessness (Other): Person in the case is a male. Symptom in the case is breathlessness.
  Interventions: Other: Person in the case is a male.; Other: Symptom in the case is breathlessness.
- Man+Pain (Other): Person in the case is a male. Symptom in the case is pain.
  Interventions: Other: Person in the case is a male.; Other: Symptom in the case is pain.
- Woman+Breathlessness (Other): Person in the case is a female. Symptom in the case is breathlessness.
  Interventions: Other: Person in the case is a female.; Other: Symptom in the case is breathlessness.
- Woman+Pain (Other): Person in the case is a female.Symptom in the case is pain.
  Interventions: Other: Person in the case is a female.; Other: Symptom in the case is pain.

INTERVENTIONS:
Other: Person in the case is a male. — Person in the case is a male.
  Arms: Man+Breathlessness; Man+Pain
Other: Person in the case is a female. — Person in the case is a female.
  Arms: Woman+Breathlessness; Woman+Pain
Other: Symptom in the case is breathlessness. — Symptom in the case is breathlessness.
  Arms: Man+Breathlessness; Woman+Breathlessness
Other: Symptom in the case is pain. — Symptom in the case is pain.
  Arms: Man+Pain; Woman+Pain

SUMMARY:
This is a web-based randomized survey to evaluate management of respiratory symptoms among physicians in Sweden. The aim of this study is to determine if there is a gender bias in the diagnosis of COPD and how often physicians identify that chronic refractory breathlessness requires treatment as compared to refractory pain.

DETAILED DESCRIPTION:
BACKGROUND:

Chronic obstructive pulmonary disease (COPD) is a major cause of morbidity and mortality worldwide. An American randomized web-based study showed important differences in the diagnosis of COPD among female and male patients.Women were more likely to be misdiagnosed as chronic cough or asthma instead of COPD and physicians were more reluctant to refer further women for spirometry.This is of importance as treatment and follow-up differ between the conditions.

Breathlessness, a subjective experience of breathing discomfort, is the cardinal symptom of cardiac and pulmonary disease. In advanced COPD, 98% of patients experience breathlessness which persists at rest or on minimal exertion, despite optimal treatment of the underlying disease (chronic refractory breathlessness). Dyspnea is linked to reduced physical activity, worsening deconditioning, increased anxiety and depression, impaired quality of life, loss of the will to live near death, increased risk of hospitalization, and earlier death.

The preferred treatment for the relief of chronic refractory breathlessness is a systemic (oral or parenteral) low dose opioid (Level I evidence). In a recent meta-analysis of 16 studies (271 patients in total), low dose opioids reduced chronic refractory breathlessness in advanced COPD, without any reported serious adverse effects. Lower dose opioids were not associated with increased risk of admission to hospital or death in a large register-based Swedish study of 2,249 patients with oxygen-dependent COPD patients treated with lower dose opioids (≤ 30mg of oral morphine/day).

Despite the growing evidence that support the use of opioids, physicians are reluctant to prescribe low dose opioids for breathlessness in COPD. In a review of 2000 random dispensed opioid prescriptions among patients with advanced COPD, most of whom suffered from severe chronic breathlessness, the most common stated indication was pain (97%), with only 2% for breathlessness. In a survey, Dutch chest physicians were reluctant to prescribe opioids for refractory breathlessness in advanced COPD due to perceived resistance from the patient and fear of adverse effects, including respiratory depression. Qualitative studies from Canada has shown that physicians in pulmonary medicine and primary care, families and patients feel that low dose opioids can be helpful for the relief of breathlessness, but that treatment was delayed or avoided due to lack of guidelines, lack of related knowledge and experience about opioids, and fears related to the potential adverse effects and legal censure.

No randomized trial has compared how physicians assess and treat refractory breathlessness versus refractory pain, how often opioids are considered for treatment of breathlessness and what factors affect the choice of treatment in chronic breathlessness as compared to pain in advanced COPD. Furthermore, it remains unknown if there is a gender bias in the diagnosis of COPD among physicians treating COPD patients.

METHOD:

This is a randomized, triple-blind, parallel group-, web-based study based on a survey instrument which is answered by certified physicians who treat patients with respiratory problems in Sweden. The survey is based upon a hypothetical patient case which regards situations and considerations that are part of physicians' daily clinical management and treatment of COPD patients. Two randomizations take place regarding the hypothetical case 1) Sex 2) Symptom. The participant is shown a hypothetical patient case which is randomized (1:1:1:1) regarding sex and symptom to one of four potential case scenarios: man+breathlessness; man+pain; woman+breathlessness; or woman+pain.

AIM:

The aim of the study is to determine if there is a gender bias in the diagnosis of COPD; how often physicians identify that chronic refractory breathlessness requires treatment as compared to refractory pain, which symptomatic treatments are considered with focus on morphine; explore physicians perception regarding the grade of evidence for different treatments for the relief of chronic breathlessness; and examine which factors affect physicians decision to treat refractory breathlessness with opioids.

ELIGIBILITY:
Inclusion Criteria (all required):

* Certified physician
* Treats patients with respiratory symptoms and reduced physical activity
* Able to read and understand a hypothetical case in Swedish

Exclusion Criteria:

* Knowledge about the aim and/or design of the study, or
* Previous participation in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
COPD treatment in the Questionnaire | through study completion, up to 6 months
  Would there be a difference between the hypothetical case with breathlessness compared to the otherwise identical case with pain instead of breathlessness regarding:
  1. Proportion of study participants that consider that the patient in the case is not optimally treated;
  2. Proportion of study participants that consider morphine as either primary or secondary treatment option

SECONDARY OUTCOMES:
Gender bias in COPD diagnosis in the Questionnaire | through study completion, up to 6 months
  Would there be a difference between the cases with a male respective female patient regarding:
  * Proportion of study participants that consider COPD diagnosis;
  * Proportion of study participants that consider spirometry for further diagnostics
Symptomatic treatment in the Questionnaire | through study completion, up to 6 months
  Would there be a difference between the case with breathlessness compared with the case with pain regarding:
  * Chosen treatment options;
  * Reasons not to choose treatment with opioids Chosen treatment options Reasons not to choose treatment with opioids

OTHER OUTCOMES:
Non-randomized measurements in the Questionnaire | through study completion, up to 6 months
  Proportion of study participants that consider the described breathlessness to be refractory
Chosen evidence-grades as non-randomized measurements in the Questionnaire | through study completion, up to 6 months
  Chosen evidence-grades for treatment options of refractory breathlessness
Chosen potential risks as non-randomized measurements in the Questionnaire | through study completion, up to 6 months
  Chosen potential risks with opioid treatment

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Ekström, MD, PhD, Principal Investigator — Department of Medicine, Blekinge Hospital, SE-37185 Karlskrona
Locations (1):
- Department of Respiratory Medicine and Allergology, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmadi Z, Sandberg J, Shannon-Honson A, Vandersman Z, Currow DC, Ekstrom M. Is chronic breathlessness less recognised and treated compared with chronic pain? A case-based randomised controlled trial. Eur Respir J. 2018 Sep 15;52(3):1800887. doi: 10.1183/13993003.00887-2018. Print 2018 Sep. PMID 30002106